CLINICAL TRIAL: NCT04493268
Title: HYPONATREMIA AND INFLAMMATION AND CLINICAL OUTCOMES IN HOSPITALIZED COVID-19 PATIENTS
Brief Title: HYPONATREMIA IN COVID-19 PATIENTS
Status: Completed | Type: Observational
Sponsor: Hospital Nacional Profesor Alejandro Posadas (Other)
Responsible Party: Principal Investigator, Ladislao Diaz Ballve, GRADUATE IN KINESIOLOGY, Hospital Nacional Profesor Alejandro Posadas
Other Study IDs: HYPONATREMIA IN COVID PATIENTS
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Hyponatremia; Covid19; Corona Virus Infection
Keywords: INFLAMMATION; COVID; CORONA
MeSH Terms: conditions — Hyponatremia; COVID-19; Coronavirus Infections; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SYSTEMIC INFLAMMATION HAS BEEN ASSOCIATED WITH SEVERE COVID-19. HYPONATREMIA CAN RESULT FROM INFLAMMATION DUE TO NON-OSMOTIC STIMULI FOR VASOPRESSIN PRODUCTION. IN THIS PROSPECTIVE COHORT STUDY WE ANALIZED DATA FROM PATIENTS WITH COVID-19 AND THE ASOCIATION WITH HYPONATREMIA AND CLINICAL OUTCOMES.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS WITH SARS-CoV-2 INFECTION CONFIRMED BY PCR OF NASOPHARYNGEAL SWABS.

Exclusion Criteria:

-

Ages: 1 Month to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: GENERAL POPULATION
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-03-07 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
MORTALITY | 30 DAYS
  HYPONATREMIA AND MORTALITY

SECONDARY OUTCOMES:
ICU HOSPITALIZATION | 30 DAYS
  HYPONATREMIA AND ICU HOSPITALIZATION

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS EGHI, physician, Principal Investigator — University of Buenos Aires
Locations (1):
- Hospital Posadas, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ayus JC, Negri AL, Moritz ML, Lee KM, Caputo D, Borda ME, Go AS, Eghi C. Hyponatremia, Inflammation at Admission, and Mortality in Hospitalized COVID-19 Patients: A Prospective Cohort Study. Front Med (Lausanne). 2021 Dec 2;8:748364. doi: 10.3389/fmed.2021.748364. eCollection 2021. PMID 34926496